CLINICAL TRIAL: NCT04510519
Title: Scaling Mental Healthcare in COVID-19 With Voice Biomarkers: An Observational Study
Brief Title: Scaling Mental Healthcare in COVID-19 With Voice Biomarkers
Status: Completed | Type: Observational
Sponsor: Kintsugi Mindful Wellness, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: COV-1
Record Dates: First submitted 2020-08-07; First posted 2020-08-12 (Actual); Last update posted 2022-09-30 (Actual); Status verified 2022-09

CONDITIONS: Major Depressive Disorder; Generalized Anxiety
MeSH Terms: conditions — Depressive Disorder, Major; Generalized Anxiety Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to advance research on group sessions for mental health. The first-of-its-kind study measuring various features in a group setting, combining rich metadata in creating state-of-the-art machine learning models, and developing workflows for mental health that are both scalable and personalized.

DETAILED DESCRIPTION:
The anticipated impact of this study is defining voice biomarker features and reward functions for a deep reinforcement learning based system from group interactions that improve depression and anxiety outcomes. The investigators' ability to quantify the real-time impact of human-intervention in scaled group video sessions can be very meaningful for creating best practices in the area where measurement is infrequent.

The investigators' priority is to scale the optimal mix of individuals for group therapy sessions based on reward functions that maximize improvements in depression and anxiety scores. Current group therapy appointments may track little save few who use various group feedback questionnaires (e.g. OQ, GCQ, or GQ). Voice biomarkers can play a key role in the real-time measurement of mental health.

The proposed work is to conduct a feasibility study on creating reward functions that most effectively enable engagement for group sessions as measured by voice biomarkers before, during, and after group video meetings.

ELIGIBILITY:
Inclusion Criteria:

* Ownership of a personal iPhone (version iOS 12.0 or later) and willingness to install and maintain the Kintsugi app for remote participation throughout the study duration
* Able to understand and comply with instructions in English

Exclusion Criteria:

* Has any other clinically significant medical condition or circumstance that, in the opinion of the Investigator, could affect patient safety, preclude evaluation of response, interfere with the ability to comply with study procedures, or prohibit completion of the study
* Has a visual or physical motor impairment that could interfere with study tasks
* Is site personnel directly affiliated with this study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes men and women over the age of 18 years
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | March 30, 2021
  A repeated measures, within-subject design using exploratory techniques will identify the best group session features or combination of features that correlate with or predict change on the PHQ-9.
Generalized Anxiety Disorder (GAD-7) | June 20, 2021
  A repeated measures, within-subject design using exploratory techniques will identify the best group session features or combination of features that correlate with or predict change on the GAD-7.

CONTACTS AND LOCATIONS:
Locations (1):
- Kintsugi Mindful Wellness, Inc., Berkeley, California, United States